CLINICAL TRIAL: NCT02034526
Title: A Randomised Controlled Trial of Reducing Atrial Pacing Rate to Reduce Atrial Fibrillation in Patients With Sick Sinus Syndrome and Dual Chamber Pacemaker.
Brief Title: Reducing Atrial Pacing Rate to Reduce Atrial Fibrillation in Patients With Sick Sinus Syndrome.
Acronym: DANPACEII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Herning Hospital (Other); Regionshospitalet Viborg, Skive (Other); Aabenraa Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Vejle Hospital (Other); Odense University Hospital (Other); Zealand University Hospital (Other); Rigshospitalet, Denmark (Other); Bispebjerg Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Jens Cosedis Nielsen, Jens Cosedis Nielsen, professor, MD, DMSc, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-2013-225-13
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Sinus Node Disease; Atrial Fibrillation
Keywords: Sinus node disease; Atrial fibrillation; Pacing
MeSH Terms: conditions — Sick Sinus Syndrome; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DDDR-60 (Placebo Comparator): DDDR, lower pacing rate 60 bpm, RR activated (low-moderate)
  Interventions: Device: DDDR-60
- DDD-40 (Experimental): DDD, lower pacing rate 40 bpm, RR function off
  Interventions: Device: DDD-40

INTERVENTIONS:
Device: DDDR-60 — DDDR, lower pacing rate 60 bpm, RR activated (low-moderate)
  Arms: DDDR-60
Device: DDD-40 — DDD, lower pacing rate 40 bpm, RR function off
  Arms: DDD-40

SUMMARY:
Atrial fibrillation (AF) is prevalent in patients with sick sinus syndrome (SSS) and associated with an increased risk of stroke and death. Within the first two years after pacemaker implantation almost half of the patients are diagnosed with AF. Studies have indicated that an increased amount of stimulation from the pacemaker in the atria is associated with an increased amount of AF.

The aim of the present study is to test the hypothesis that a reduction of stimulation from the pacemaker in the atria, and reducing the minimal heart rate, increases the time to AF.

ELIGIBILITY:
Inclusion Criteria:

* Sick sinus syndrome with and without AV block and indication for first-time implantation of a DDD pacemaker: symptomatic sinus pauses (>2 sec) or bradycardia with or without paroxysmal AF.
* Age ≥18 years.
* Patient informed consent.

Exclusion Criteria:

* Permanent or persisting (>7 days) AF prior to implantation.
* Persisting symptomatic sinus bradycardia and/or chronotropic incompetence where DDD-pacing at a frequency of >40 bpm is indicated (verified with long term ECG monitoring).
* Life expectancy <2 years.
* Participation in another interventional research study.
* Indication for implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT).
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2014-05; Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Time to first episode of AF>6 min detected by the pacemaker | Within two years
  First episode of AF > 6 min detected by the device

SECONDARY OUTCOMES:
Time to first episode of AF>6 hours detected by the pacemaker | Within two years
  First episode of AF > 6 hours detected by the device
Time to first episode of AF>24 hours detected by the pacemaker | Within two years
  First episode of AF > 24 hours detected by the device
Time to direct current (DC) cardioversion or medical cardioversion for AF | Within two years
  Time to direct current (DC) cardioversion or medical cardioversion for AF
Time to stroke, transient ischemic attack (TIA), or thromboembolic event | Within two years
  Time to stroke, transient ischemic attack (TIA), or thromboembolic event
Time to death | Within two years
  Time to all cause death
QOL | After 12 months
  Quality of life assessment with SF-36
6MHWT | After 12 months
  6-minute hall walk test
Time to need for reprogramming of the pacing rate (cross-over) | Within 2 years
  Time to need for reprogramming of the pacing rate (cross-over)

CONTACTS AND LOCATIONS:
Overall Officials: Jens C Nielsen, prof., DMSc,, Principal Investigator — Department of Cardiology, Aarhus University Hospital
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Aarhus N, Denmark

REFERENCES:
- [Derived] Kronborg MB, Frausing MHJP, Malczynski J, Riahi S, Haarbo J, Holm KF, Larroude CE, Albertsen AE, Svendstrup L, Hintze U, Pedersen OD, Davidsen U, Fischer T, Johansen JB, Kristensen J, Gerdes C, Nielsen JC; DANPACE II Investigators. Atrial pacing minimization in sinus node dysfunction and risk of incident atrial fibrillation: a randomized trial. Eur Heart J. 2023 Oct 21;44(40):4246-4255. doi: 10.1093/eurheartj/ehad564. PMID 37638973

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT02034526/Prot_SAP_000.pdf